CLINICAL TRIAL: NCT02662985
Title: A 52-week, Multicenter Study to Assess the Time Course of Response to Secukinumab on Joint Inflammation Using Power Doppler Ultrasonography in Patients With Active Psoriatic Arthritis
Brief Title: Study of Power Doppler Ultrasound (PDUS) to Measure Response of Secukinumab Treatment in Patients With Active Psoriatic Arthritis (PsA)
Acronym: PDUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457F2354; 2015-002394-38 (EudraCT Number)
Record Dates: First submitted 2016-01-13; First posted 2016-01-26 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Psoriatic Arthritis
Keywords: Power Doppler Ultrasonography; Psoriatic Arthritis; Enthesitis; Synovitis; Outcome Measures in Rheumatology; Spondyloarthritis Research Consortium of Canada; active psoriatic arthritis; secukinumab; Arthritis; GLOESS; monoclonal antibody; PsA
MeSH Terms: conditions — Arthritis, Psoriatic; Synovitis; Arthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): In Treatment Period-1:
  Patients in this group were administered secukinumab with 12 weeks of treatment from baseline.
  In Treatment Period-2:
  Patients continued to receive the same active dose of secukinumab every 4 weeks until Week 24
  In Treatment Period 3 (extension period):
  the extension period allowed responder patients the possibility to continue open-label secukinumab treatment up to Week 52
  Interventions: Drug: AIN457 (secukinumab)
- Group 2 (Placebo Comparator): In Treatment Period-1:
  Patients received placebo at baseline and same time points as secukinumab until Week 8.
  In Treatment Period-2:
  Patients commenced open-label secukinumab every 4 weeks from Week 12, as follows, based on their clinical characteristics at Week 12
  In Treatment Period-3:
  Open-label secukinumab continued to be assigned to patients
  Interventions: Drug: AIN457 (secukinumab); Drug: Placebo

INTERVENTIONS:
Drug: AIN457 (secukinumab) — Is a recombinant monoclonal antibody which neutralizes the activity of IL-17A, and has been shown to be effective in treating patients with moderate-to-severe plaque psoriasis.
  Secukinumab 150 mg provided in 1 mL pre filled syringes (PFS) for s.c. injection. The 300 mg dose was administered as 2 × PFS injections.
  Other Names: Secukinumab
Drug: Placebo — Secukinumab placebo was provided in a 1 mL PFS for s.c. injection.
  Arms: Group 2

SUMMARY:
This study was designed to leverage the sensitivity of ultrasonography available in clinical practice setting to better describe the time course of response to secukinumab (150 mg and 300 mg) on joint synovitis and enthesitis in PsA patients with an inadequate response to non-biologic DMARDs. PDUS changes in joint synovitis will be assessed using the global Outcome Measures in Rheumatology (OMERACT)-European League against Rheumatism (EULAR) synovitis score (GLOESS) and changes in joint enthesitis were assessed using the OMERACT enthesitis score.

DETAILED DESCRIPTION:
This was a 52-week, multicenter, international study consisting of a 2 to 4-week Screening period, a 12-week randomized, placebo-controlled double-blind treatment period (Period 1), a 12-week open-label treatment period (Period 2) and a 6-month open-label extension period (Period 3).

Treatment Period 1 is a 12-week placebo-controlled, randomized period primarily designed to demonstrate the early and optimal efficacy of secukinumab vs placebo on joint synovitis using PDUS via the GLOESS and global entheseal score after 12 weeks of treatment.

The main aim of Period 2 was to assess the maintenance or increased magnitude of treatment response on joint synovitis for patients from the original secukinumab groups and to assess the time course of response with secukinumab on joint synovitis in the original placebo group switched to secukinumab from Week 12.

The main aim of Period 3 (extension period) was to allow patients who respond to secukinumab to extend study treatment up to Week 52 or until commercial drug becomes available, whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand and communicate with the Investigator and comply with the requirements of the study and must provide written, signed and dated informed consent before any study assessment is performed.
2. Male or female patients at least 18 years of age.
3. Diagnosis of PsA as per CASPAR with active PsA for at least 6 months and a TJC ≥ 3 of 78 and SJC ≥ 3 of 76 at Baseline.
4. Patients must have a total synovitis PDUS score ≥ 2 and inflammation related to PD signal ≥ 1 for at least 2 (affected joints as observed via PDUS) of 48 joints at the Screening visit and at the Baseline visit (before infusion).
5. At least 1 clinically-involved enthesitis site at Screening and at the Baseline visit (before infusion) defined by SPARCC index different from 0.

Exclusion Criteria:

1. Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process obtained within 3 months prior to Screening and evaluated by a qualified physician.
2. Previous exposure to secukinumab or other biologic drug directly targeting IL-17 or IL-17 receptor.
3. Any change in the dose of oral corticosteroids in the last 4 weeks prior to the Baseline visit or use of i.v. intramuscular or intra-articular corticosteroid during the last 4 weeks prior to the enrollment visit.
4. Patients who have previously been treated with TNFα inhibitors (investigational or approved).
5. History of hypersensitivity to the study drug or its excipients or to drugs of similar classes.
6. Previous treatment with any cell-depleting therapies including but not limited to anti CD20 investigational agents (e.g. CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti CD19).
7. Prohibited psoriasis treatments/medications with topical corticosteroids in the last 4 weeks prior to randomization.
8. Pregnant or nursing (lactating) women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (4):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Wheaton, Maryland
  - Novartis Investigative Site, Salt Lake City, Utah
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, San Miguel de Tucumán
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Bogota, Cundinamarca, Colombia
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- France (3):
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
- Novartis Investigative Site, Miskolc, Baz, Hungary
- Novartis Investigative Site, Dublin, Ireland
- Italy (3):
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Pisa
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Guadalajara Jalisco, Mexico
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] D'Agostino MA, Schett G, Lopez-Rdz A, Senolt L, Fazekas K, Burgos-Vargas R, Maldonado-Cocco J, Naredo E, Carron P, Duggan AM, Goyanka P, Boers M, Gaillez C. Response to secukinumab on synovitis using Power Doppler ultrasound in psoriatic arthritis: 12-week results from a phase III study, ULTIMATE. Rheumatology (Oxford). 2022 May 5;61(5):1867-1876. doi: 10.1093/rheumatology/keab628. PMID 34528079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 166 participants enrolled in 17 countries
Pre-assignment Details: 83 partcipants were randomized to each group
Groups:
- Group 1 - Secukinumab (150 mg + 300 mg): In Treatment Period-1:
  Patients in this group were administered secukinumab with 12 weeks of treatment from baseline.
  In Treatment Period-2:
  Patients continued to receive the same active dose of secukinumab every 4 weeks until Week 24 (although primary outcome was to week 12 only)
  In Treatment Period 3 (extension period):
  the extension period allowed responder patients the possibility to continue open-label secukinumab treatment up to Week 52
- Group 2 - Placebo/Secukinumab: In Treatment Period-1:
  Patients received placebo at baseline and same time points as secukinumab until Week 8.
  In Treatment Period-2:
  Patients commenced open-label 150 or 300 mg secukinumab every 4 weeks from Week 12, as follows, based on their severity of skin disease at Week 12
  In Treatment Period-3:
  Open-label secukinumab continued to be assigned to patients
Period: Treatment Period 1
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Started | 83 | 83
Completed | 82 | 79
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Started | 82 | 79
Completed | 81 | 78
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Treatment Period 3 (Extension Period)
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Started | 81 | 78
Completed | 75 | 69
Not Completed | 6 | 9
Not completed — Withdrew before entering period | 4 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 2 - Placebo/Secukinumab (150 mg + 300 mg): In Treatment Period-1:
  Patients received placebo at baseline and same time points as secukinumab until Week 8.
  In Treatment Period-2:
  Patients commenced open-label secukinumab 150 or 300 mg every 4 weeks from Week 12, as follows, based on their severity of skin disease at Week 12
  In Treatment Period-3:
  Open-label secukinumab continued to be assigned to patients
- Total: Total of all reporting groups
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab (150 mg + 300 mg) | Total
Number analyzed (Participants) | 83 | 83 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 79 | 155
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (12.35) | 46.7 (12.08) | 46.7 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 38 | 37 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 75 | 75 | 150
  Asian | 1 | 0 | 1
  Native American | 4 | 8 | 12
  Unknown | 2 | 0 | 2
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Secukinumab and Placebo in Terms of Joint Synovitis as Measured by the Power Doppler Ultrasonography (PDUS) Global OMERACT-EULAR Synovitis Score (GLOESS)
Description: Mixed model repeated measures (MMRM) analysis of change in Global OMERACT-EULAR Synovitis Score (GLOESS) score at Week 12 (observed data) to compare treatments
  The range for the GLOESS score is 0 to 144. GLOESS is the ultrasound scoring system measured for 24 pairs of joints. The scoring is from 0 to 3 for each joint; so the minimum score can be 0 and maximum can be 144.
Time Frame: 12 weeks
Population: Full analysis set (FAS): The FAS comprised all patients from the Randomized set to whom study treatment had been assigned. Following the intent-to-treat principle, patients were analyzed according to the treatment assigned at randomization.
Measure: Mean (Standard Error); unit: Adjusted Mean Change in scores
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Number analyzed (Participants) | 83 | 81
Adjusted Mean Change in scores | -9.05 (0.94) | -5.86 (0.93)
Statistical Analysis 1: Comparison: Group 1 - Secukinumab (150 mg + 300 mg) vs Group 2 - Placebo/Secukinumab; GLOESS scores; Test type: Superiority; p = 0.0040, Mixed Models Analysis; mixed model repeated measures (MMRM); Median Difference (Net) = -3.18, 95% CI 2-sided [-5.52 to -0.85], Standard Error of Mean 1.18

2. Secondary Outcome: Proportion of Participants With American College of Rheumatology (ACR)-20 Response
Description: ACR 20 responder has ≥ 20% improvement in TJC and SJC and >20% improvement in 3 of the following 5 domains: patient's assessment of disease activity, physician's assessment of disease activity, patient's
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Number analyzed (Participants) | 83 | 83
Participants | 56 | 26
Statistical Analysis 1: Comparison: Group 1 - Secukinumab (150 mg + 300 mg) vs Group 2 - Placebo/Secukinumab; Proportion of patients with ACR 20 response at Week 12 (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; Logistic regression using non-responder imputation; Odds Ratio (OR) = 4.60, 95% CI 2-sided [2.38 to 8.89]

3. Secondary Outcome: Proportion of Participants With American College of Rheumatology (ACR)-50 Response
Description: ACR 50 responder has ≥ 50% improvement in TJC and SJC and >25% improvement in 3 of the following 5 domains: patient's assessment of disease activity, physician's assessment of disease activity, patient's assessment of PsA pain, HAQ-DI, or hsCRP.
Time Frame: Week 12
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Number analyzed (Participants) | 83 | 83
Participants | 38 | 7
Statistical Analysis 1: Comparison: Group 1 - Secukinumab (150 mg + 300 mg) vs Group 2 - Placebo/Secukinumab; Proportion of patients with ACR 50 response at Week 12 (FAS); Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 9.65, 95% CI 2-sided [3.92 to 23.75]

4. Secondary Outcome: Spondyloarthritis Research Consortium of Canada (SPARCC)
Description: Repeated measures mixed effect (MMRM) analysis of SPARCC total score change from baseline to Week 12 between the 2 treatment groups.
  SPARCC index ranges from 0 to 16.
Time Frame: Baseline to Week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Error); unit: Adjusted mean change in scores
Arm/Group | Group 1 - Secukinumab (150 mg + 300 mg) | Group 2 - Placebo/Secukinumab
Number analyzed (Participants) | 83 | 81
Adjusted mean change in scores | -2.23 (0.29) | -1.57 (0.29)
Statistical Analysis 1: Comparison: Group 1 - Secukinumab (150 mg + 300 mg) vs Group 2 - Placebo/Secukinumab; SPARCC; Test type: Superiority; p = 0.0327, Regression, Logistic; Adjusted mean of treatment difference = -0.67, 95% CI 2-sided [-1.374 to 0.043], Standard Error of Mean 0.36

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for 12 weeks. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 52 weeks
Description: Adverse Events (AEs) are any untoward sign or symptom that occurs during the study treatment period
Groups:
- Treatment Group 1 - Secukinumab (150+300 mg): In Treatment Period-1:
  Patients in this group were administered secukinumab with 12 weeks of treatment from baseline.
  In Treatment Period-2:
  Patients continued to receive the same active dose of secukinumab every 4 weeks until Week 24 (although primary outcome was to week 12 only)
  In Treatment Period 3 (extension period):
  the extension period allowed responder patients the possibility to continue open-label secukinumab treatment up to Week 52
- Treatnent Group 2 - Placebo/Secukinumab: In Treatment Period-1:
  Patients received placebo at baseline and same time points as secukinumab until Week 8.
  In Treatment Period-2:
  Patients commenced open-label 150 or 300 mg secukinumab every 4 weeks from Week 12, as follows, based on their severity of skin disease at Week 12
  In Treatment Period-3:
  Open-label secukinumab continued to be assigned to patients
Arm/Group | Treatment Group 1 - Secukinumab (150+300 mg) | Treatnent Group 2 - Placebo/Secukinumab
All-Cause Mortality (participants affected / at risk) | 1/161 | 0/83
Serious Adverse Events (participants affected / at risk) | 9/161 | 2/83
Other Adverse Events (participants affected / at risk) | 79/161 | 27/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 - Secukinumab (150+300 mg) (N=161) | Treatnent Group 2 - Placebo/Secukinumab (N=83)
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 - Secukinumab (150+300 mg) (N=161) | Treatnent Group 2 - Placebo/Secukinumab (N=83)
Dry eye (Eye disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Constipation (Gastrointestinal disorders) | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 4 | 1
Fatigue (General disorders) | 4 | 0
Bronchitis (Infections and infestations) | 8 | 2
Gastroenteritis (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 7 | 3
Nasopharyngitis (Infections and infestations) | 19 | 4
Oral herpes (Infections and infestations) | 4 | 1
Pharyngitis (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Urinary tract infection (Infections and infestations) | 10 | 3
Fall (Injury, poisoning and procedural complications) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 13 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypertension (Vascular disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT02662985/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/85/NCT02662985/SAP_001.pdf